CLINICAL TRIAL: NCT03877614
Title: Application of Artificial Intelligence Deep Learning to the Correlation Between Cardiovascular Disease and Individualized Differences
Brief Title: Artificial Intelligence With Deep Learning and Genes on Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ping-Yen Liu, Director of Cardiology, Internal Medicine and Professor of Institute of Clinical Medicine, National Cheng-Kung University Hospital
Other Study IDs: A-ER-107-149
Record Dates: First submitted 2019-03-08; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary DNA with genetic polymorphism chips comparative analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiovascular high-risk (disease) group: A. Coronary artery disease B. Congestive heart failure with reduced ejection fraction C. Hypertrophic cardiomyopathy D. Atrial fibrillation E. Pulmonary hypertension F. Fabry's disease
  Interventions: Other: ASCVD risk score
- Cardiovascular Low-risk (control) group: Patient with only risk factors with ASCVD score<10% will be recognized as the comparison group
  Interventions: Other: ASCVD risk score

INTERVENTIONS:
Other: ASCVD risk score — ASCVD score< 10% will be in the control or low-risk group

SUMMARY:
An association study with large database from electronic medical record system, images, outcome analysis and genetic single nucleotide polymorphism variations by machine learning and artificial intelligence methods in a Taiwanese and Chinese medical center based population

DETAILED DESCRIPTION:
In recent years, the analysis of big data database combined with computer deep learning has gradually played an important role in biomedical technology. For a large number of medical record data analysis, image analysis, single nucleotide polymorphism difference analysis, etc., all relevant research on the development and application of artificial intelligence can be observed extensively. For clinical indication, patients may receive a variety of cardiovascular routine examination and treatments, such as: cardiac ultrasound, multi-path ECG, cardiovascular and peripheral angiography, intravascular ultrasound and optical coherence tomography, electrical physiology, etc... The current study is for the investigative cardiovascular team to take the advantage that in addition to the examination and treatment the participants should appropriately receive, the investigators can also analyze the individual differences and using the "deep learning methodology" to analyze the difference in physical fitness, therapeutic effectiveness and the consideration in the safety of the treatment. The additional goal of this study is to improve the quality of health care, the realization of cardiovascular "precise medicine" especially with personal difference on genetic variation.

This study will analyze the differences in the individualization of cardiovascular disease between diseases and other subjects to further improve the quality of care for clinical patients. By using artificial intelligence deep learning system, the investigators hope to not only improve the diagnostic rate and also gain more accurately predict the patient's recovery, improve medical quality in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Patients' selection criteria and enrollment plan:

We will enroll subjects from either cardiovascular clinics or inpatients from the National Cheng Kung University Hospital from 2018 to 2021 after the signature of inform consent from patients and their families. The major enrollment criteria include one of the flowing diseases or conditions:

A. Coronary artery disease:

1. History of myocardial infarction
2. Coronary artery disease with computer tomography angiography image study with at least one vessel luminal stenosis >70%
3. Coronary artery stents implantation by hospital-based image database
4. Thallium-201 scan positive/treadmill test positive with additional 2 risk factors, including

   1. Diabetes mellitus
   2. Hypertension
   3. Dyslipidemia
   4. Family history of sudden death, coronary bypass surgery, cerebral vascular attacks (CVA), premature myocardial infarction
   5. Smoking behaviors

B. Congestive heart failure with reduced ejection fraction

1. Echocardiography left ventricular ejection fraction <40%

C. Hypertrophic cardiomyopathy:

1. Left ventricle interventricular septum（IVS) >15 mm
2. Left ventricle mass index> 200gm
3. Apical hypertrophy noted on the report with 4 chamber view

D. Atrial fibrillation

1. Recorded by Holter continuous EKG
2. Recorded by standard 12 leads complete EKG

E. Pulmonary hypertension

1. Echo with systolic pulmonary pressure (sysPAP)> 40 mmHg
2. Diagnosis of idiopathic pulmonary hypertension
3. Under pulmonary hypertension medication

F. Fabry's disease

1. α-Galactosidase (a-GAL) enzyme deficiency
2. Genetic disorder

G. Patient with only risk factors (<3 risk factors), recognized as the comparison group (>500 cases)

1. Diabetes mellitus
2. Hypertension
3. Dyslipidemia
4. Family history of sudden death, coronary bypass surgery, cerebral vascular attacks, premature myocardial infarction
5. Smoking behavior

Exclusion Criteria:

* Patients unwilling to be enrolled
* Concentration of DNA collection was inadequate after 3 times of collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pipeline for case enrollment:
  1. We will enroll investigating subjects from the clinics of near 10 physicians screened by our assistant or physicians themselves, with nearly 100-120 cases/month. According to our initial experience during our previous hospital-based grant in 2018 showed feasible case number to be enrolled, nearly 1000 case within 3 months enrollment. In total, we plan to recruit 5000 subjects with cardiovascular disease or with risk factors within 3 years. (IRB approval A-ER-107-149)
  2. Our study subjects will be evaluated whether they fulfill the cases criteria by an independent physician every month.
  3. In comparison with disease, the risk factor only group (500 cases) will be the matching group on genetic background and outcome comparison.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular events | 5 years
  The rate of myocardial infarction, stroke, death, cardiovascular death, heart failure with hospitalization

SECONDARY OUTCOMES:
Heart function changes | 5 years
  parameters and function changes from echocardiography
Lipid profiles | 5 years
  The percentage changes and response of lipid profile with regular lipid lowering agents
Arrhythmia events | 5 years
  The rate of arrhythmia associated complications and clinical events, stokes
Recurrent acute coronary events | 5 years
  The rate of recurrent acute coronary events with hospitalization needed or re-intervention procedures for coronary artery needed

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu YL, Huang MS, Chang HY, Lee CH, Chen DP, Li YH, Chao TH, Liu YW, Liu PY. Application of genetic risk score for in-stent restenosis of second- and third-generation drug-eluting stents in geriatric patients. BMC Geriatr. 2023 Jul 19;23(1):443. doi: 10.1186/s12877-023-04103-w. PMID 37468836
- [Derived] Lee PT, Huang MH, Huang TC, Hsu CH, Lin SH, Liu PY. High Burden of Premature Ventricular Complex Increases the Risk of New-Onset Atrial Fibrillation. J Am Heart Assoc. 2023 Feb 21;12(4):e027674. doi: 10.1161/JAHA.122.027674. Epub 2023 Feb 15. PMID 36789835